CLINICAL TRIAL: NCT04370548
Title: A Phase 3 Multi-Center, Double-Blind, Placebo-Controlled, Randomized Study of DARE-BV1 in the Treatment of Bacterial Vaginosis
Brief Title: DARE-BV1 in the Treatment of Bacterial Vaginosis (DARE-BVFREE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daré Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DARE-BV1-001
Record Dates: First submitted 2020-04-03; First posted 2020-05-01 (Actual); Results first posted 2021-07-02 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly assigned to one of the following treatment groups (2:1): DARE- BV1 clindamycin phosphate vaginal gel, 2% (1 dose is 5 g gel = 100 mg clindamycin) QD × 1 day, or placebo vaginal gel (Universal HEC Placebo Gel), 5g, QD × 1 day. Study drug will be applied intravaginally within 1 day of randomization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clindamycin phosphate vaginal gel, 2% (Experimental)
  Interventions: Drug: DARE-BV1clindamycin phosphate vaginal gel, 2%
- Placebo vaginal gel (Universal HEC Placebo Gel) (Placebo Comparator)
  Interventions: Drug: DARE-BV1clindamycin phosphate vaginal gel, 2%

INTERVENTIONS:
Drug: DARE-BV1clindamycin phosphate vaginal gel, 2% — One full applicator (5 g) of clindamycin phosphate vaginal gel, 2% (100 mg clindamycin) or placebo gel will be applied intravaginally as a single dose within 1 day of randomization.
  Other Names: Placebo vaginal gel (HEC Universal Placebo Gel)

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study of DARE-BV1 (clindamycin phosphate vaginal gel, 2%) (QD x 1 day) compared to placebo vaginal gel (HEC Universal Placebo Gel) (QD × 1 day) for the treatment of bacterial vaginosis. Patients will be evaluated at three time points: a Day 1 Screening/Randomization visit, a Day 7-14 Interim Assessment visit, and a Day 21 - 30 Test of Cure [TOC] visit). Patients who discontinue prematurely from the study will receive a safety follow-up phone call between Day 21-30. The total study duration will be approximately one month for each individual patient.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must provide written informed consent prior to any study-related procedures being performed. Patients from 12 through 17 years old may participate where permitted by applicable local regulations and Institutional Review Board (IRB) approval and with appropriate documentation of consent from the parent(s)/guardian(s) and assent from the patient.
2. Participants must have a clinical diagnosis of bacterial vaginosis, defined as having all of the following:

   1. Off-white (milky or gray), thin, homogeneous discharge with minimal or absent pruritus and inflammation of the vulva and vagina
   2. The presence of clue cells > 20% of the total epithelial cells on microscopic examination of the saline wet mount
   3. Vaginal secretion pH of > 4.5
   4. A fishy odor of the vaginal discharge with the addition of a drop of 10% KOH (i.e., a positive "whiff test")
3. Participants must be females ≥ 12 years of age with no known medical conditions that, in the Investigator's opinion, may interfere with study participation.
4. Participants must agree to abstain from sexual intercourse and/or sexual activity throughout the first seven days following treatment. Patients must also agree to use adequate birth control (see Inclusion Criterion #5) should they later engage in heterosexual intercourse through the final study visit (Day 21-30).
5. Participants of childbearing potential must have a negative urine pregnancy test result at screening, should use adequate birth control after the first seven days of treatment if engaging in heterosexual intercourse, and should not plan on becoming pregnant for the duration of the study. Acceptable forms of birth control include oral contraceptives (the pill), intrauterine devices (IUDs), contraceptive implants under the skin, patches or injections, and non-polyurethane condoms (e.g., latex, polyisoprene) with or without spermicide. Patients in monogamous relationships with vasectomized males may also participate. Abstinence may be allowed, but requires Medical Monitor (or designee) approval prior to randomization. Oral or transdermal hormonal contraceptives must be in use for one full cycle (e.g., four to eight weeks) prior to study drug application. Injectable or implanted contraceptives (e.g., Depo-Provera, Nexplanon, or hormonal IUD) must be injected/inserted at least seven days prior to study drug application. Participants who are not of childbearing potential, as defined below, must also have a negative urine pregnancy test prior to randomization:

   1. Postmenopausal for at least one year prior to the Entry Visit (Visit 1) (defined as amenorrheic for more than one continuous year), or
   2. Surgically sterile (defined as bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) at least 6 months before first dose, or
6. Non-surgical permanent sterilization procedure at least 3 months prior to first dose.
7. Participants must be willing to refrain from the use of all intra-vaginal products (e.g., douches, feminine deodorant sprays, condoms, spermicides, vaginal moisturizers and lubricants, tampons, vaginal birth control rings [e.g., NuvaRing®], and diaphragms) through the first 7 days at a minimum, and ideally through Visit 3 (Day 21-30) or Study Exit/Early Discontinuation.
8. Participants must be able to read, write, and understand English.

Exclusion Criteria:

1. Patients with active vulvovaginitis or other active infectious causes of cervicitis, vaginitis, or vulvitis (e.g., candidiasis, Trichomonas vaginalis, Chlamydia trachomatis, Neisseria gonorrhoeae, or genital lesions or ulcers consistent with human papillomavirus, active Herpes simplex, syphilis, chancroid, etc.).
2. Potential participants who are pregnant or breastfeeding, or if of child-bearing potential unwilling to practice acceptable means of birth control or abstinence during the study as described above.
3. Patients with a vaginal, vulvar, or genitourinary condition that, according to the Investigator's judgement, may confound the interpretation of clinical response.
4. Patients with a history of regional enteritis, ulcerative colitis, or a history of C. difficile associated diarrhea.
5. Patients with known current drug or alcohol abuse that could impact study compliance.
6. Patients currently receiving or who have received antifungal or antimicrobial therapy (systemic or intravaginal) within 14 days of the Screening/Randomization visit.
7. Patients who have used any other investigational product within 30 days of the screening/randomization visit.
8. Patients who will undergo evaluation or treatment during the study for abnormal cytology and/or findings from high risk HPV testing and/or Pap test finding.
9. Patients with known sensitivity to clindamycin phosphate or other lincosamides or any of the inactive ingredients in the study drug.
10. Patients with a history of any severe acute or chronic medical or psychiatric condition or laboratory abnormality that could increase the risk associated with trial participation or study treatment administration or could interfere with the interpretation of trial results and, in the judgment of the Investigator, would make the patient inappropriate for entry into the trial.

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 307 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Vision Clinical Research-Tuscon, Tucson, Arizona
  - Downtown Women's Health Care, Denver, Colorado
  - New Age Medical Research Corporation, Miami, Florida
  - Precision Clinical Research, LLC, Sunrise, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - NuDirections Clinical Research, Inc., Lawrenceville, Georgia
  - Capital Health-Lawrence OB/GYN, Lawrenceville, New Jersey
  - The Center for Women's Health & Wellness, LLC, Lawrenceville, New Jersey
  - The Jackson Clinic, PA, Jackson, Tennessee
  - Eastern Virginia Medical School, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mauck C, Hillier SL, Gendreau J, Dart C, Wu H, Chavoustie S, Sorkin-Wells V, Nicholson-Uhl CS, Perez B, Jacobs M, Zack N, Friend D. Acceptability of Single-dose Clindamycin Gel for Bacterial Vaginosis: A Randomized Controlled Trial. Clin Ther. 2023 May;45(5):415-425. doi: 10.1016/j.clinthera.2023.04.001. Epub 2023 Apr 23. PMID 37098453
- [Derived] Mauck C, Hillier SL, Gendreau J, Dart C, Chavoustie S, Sorkin-Wells V, Nicholson-Uhl C, Perez B, Jacobs M, Zack N, Friend D. Single-Dose, Bioadhesive Clindamycin 2% Gel for Bacterial Vaginosis: A Randomized Controlled Trial. Obstet Gynecol. 2022 Jun 1;139(6):1092-1102. doi: 10.1097/AOG.0000000000004805. Epub 2022 May 2. PMID 35675606

RESULTS

PARTICIPANT FLOW:
Groups:
- Clindamycin Phosphate Vaginal Gel, 2%: One full applicator (5 g) of clindamycin phosphate vaginal gel, 2% (100 mg clindamycin) will be applied intravaginally as a single dose within 1 day of randomization.
- Placebo Vaginal Gel (Universal HEC Placebo Gel): One full applicator (5 g) of placebo gel will be applied intravaginally as a single dose within 1 day of randomization.
Period: Overall Study
Arm/Group | Clindamycin Phosphate Vaginal Gel, 2% | Placebo Vaginal Gel (Universal HEC Placebo Gel)
Started | 204 | 103
Completed | 190 | 100
Not Completed | 14 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clindamycin Phosphate Vaginal Gel, 2% | Placebo Vaginal Gel (Universal HEC Placebo Gel) | Total
Number analyzed (Participants) | 204 | 103 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (8.79) | 35.2 (8.96) | 34.8 (8.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204 | 103 | 307
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 57 | 21 | 78
  Not Hispanic or Latino | 146 | 82 | 228
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 116 | 56 | 172
  White | 82 | 44 | 126
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 204 | 103 | 307
BMI, Continuous [Mean (Standard Deviation); unit: kg/m^2] | 31.75 (8.667) | 30.84 (8.183) | 31.45 (8.505)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Clinical Cure at the TOC Visit (Day 21-30).
Description: Clinical cure is defined as:
  * Resolution of the abnormal vaginal discharge associated with BV;
  * Negative 10% KOH "whiff test;" and
  * Clue cells < 20% of the total epithelial cells in the saline wet mount.
Time Frame: Visit 3 Day 21-30 post randomization
Population: Clinical Cure of the mITT Population (missing data were treated as Treatment Failure)
Measure: Count of Participants; unit: Participants
Arm/Group | Clindamycin Phosphate Vaginal Gel, 2% | Placebo Vaginal Gel (Universal HEC Placebo Gel)
Number analyzed (Participants) | 122 | 59
Participants | 86 | 21

2. Secondary Outcome: Number of Patients With Clinical Cure at the Interim Assessment Visit (Day 7-14).
Time Frame: Visit 2 Day 7-14 post randomization
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Clindamycin Phosphate Vaginal Gel, 2% | Placebo Vaginal Gel (Universal HEC Placebo Gel)
Number analyzed (Participants) | 122 | 59
Participants | 93 | 14

3. Secondary Outcome: Number of Patients With Bacteriological Cure at the TOC Visit (Day 21-30).
Description: Bacteriological cure is defined as a Nugent score < 4
Time Frame: Visit 3 Day 21-30 post randomization
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Clindamycin Phosphate Vaginal Gel, 2% | Placebo Vaginal Gel (Universal HEC Placebo Gel)
Number analyzed (Participants) | 122 | 59
Participants | 53 | 3

4. Secondary Outcome: Number of Patients With Bacteriological Cure at Interim Assessment Visit, Day 7-14
Time Frame: Visit 2, Days 7-14 post randomization
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Clindamycin Phosphate Vaginal Gel, 2% | Placebo Vaginal Gel (Universal HEC Placebo Gel)
Number analyzed (Participants) | 122 | 59
Participants | 50 | 2

5. Secondary Outcome: Number of Patients With Therapeutic Cure at the TOC Visit (Day 21-30).
Time Frame: Visit 3 Day 21-30 post randomization
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Clindamycin Phosphate Vaginal Gel, 2% | Placebo Vaginal Gel (Universal HEC Placebo Gel)
Number analyzed (Participants) | 122 | 59
Participants | 45 | 3

6. Secondary Outcome: Number of Patients With Therapeutic Cure at the Interim Assessment Visit (Day 7-14).
Time Frame: Visit 2 Day 7-14 post randomization
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Clindamycin Phosphate Vaginal Gel, 2% | Placebo Vaginal Gel (Universal HEC Placebo Gel)
Number analyzed (Participants) | 122 | 59
Participants | 43 | 0

7. Other Pre Specified Outcome: Number of Patients With Clinical Cure at the Test of Cure Visit (21-30)
Time Frame: Visit 3, Days 21-30 post randomization
Population: Per Protocol (PP) Population
Measure: Count of Participants; unit: Participants
Arm/Group | Clindamycin Phosphate Vaginal Gel, 2% | Placebo Vaginal Gel (Universal HEC Placebo Gel)
Number analyzed (Participants) | 102 | 47
Participants | 79 | 20

8. Other Pre Specified Outcome: Number of Patients With Clinical Cure at Interim Assessment Visit, Days 7-14, PP Population
Time Frame: Visit 2, Days 7-14 post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Clindamycin Phosphate Vaginal Gel, 2% | Placebo Vaginal Gel (Universal HEC Placebo Gel)
Number analyzed (Participants) | 102 | 47
Participants | 83 | 14

9. Other Pre Specified Outcome: Number of Patients With Bacteriological Cure at Test of Cure Visit, Days 21-30, PP Population
Time Frame: Visit 3, Days 21-30 post randomization
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Clindamycin Phosphate Vaginal Gel, 2% | Placebo Vaginal Gel (Universal HEC Placebo Gel)
Number analyzed (Participants) | 102 | 47
Participants | 46 | 3

10. Other Pre Specified Outcome: Number of Patients With Bacteriological Cure, Interim Assessment Visit, Days 7-14, PP Population
Time Frame: Visit 2, Days 7-14 post randomization
Population: PP Population
Measure: Count of Participants; unit: Participants
Arm/Group | Clindamycin Phosphate Vaginal Gel, 2% | Placebo Vaginal Gel (Universal HEC Placebo Gel)
Number analyzed (Participants) | 102 | 47
Participants | 45 | 1

11. Other Pre Specified Outcome: Number of Patients With Therapeutic Cure at Test of Cure Visit, Days 21-30; PP Population
Time Frame: Visit 3, Days 21-30 post randomization
Population: PP Population
Measure: Count of Participants; unit: Participants
Arm/Group | Clindamycin Phosphate Vaginal Gel, 2% | Placebo Vaginal Gel (Universal HEC Placebo Gel)
Number analyzed (Participants) | 102 | 47
Participants | 41 | 3

12. Other Pre Specified Outcome: Number of Patients With Therapeutic Cure, Interim Assessment Visit, Days 7-14, PP Population
Time Frame: Visit 2, Days 7-14 post randomization
Population: PP Population
Measure: Count of Participants; unit: Participants
Arm/Group | Clindamycin Phosphate Vaginal Gel, 2% | Placebo Vaginal Gel (Universal HEC Placebo Gel)
Number analyzed (Participants) | 102 | 47
Participants | 39 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for the entire study duration, approximately 3.5 months.
Description: There was one subject in the Clindamycin Phosphate Vaginal Gel, 2% group that withdrew from the study after randomization, but prior to dosing. This subject was not included in the safety population.
Arm/Group | Clindamycin Phosphate Vaginal Gel, 2% | Placebo Vaginal Gel (Universal HEC Placebo Gel)
All-Cause Mortality (participants affected / at risk) | 0/203 | 0/103
Serious Adverse Events (participants affected / at risk) | 0/203 | 1/103
Other Adverse Events (participants affected / at risk) | 76/203 | 28/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clindamycin Phosphate Vaginal Gel, 2% (N=203) | Placebo Vaginal Gel (Universal HEC Placebo Gel) (N=103)
Cervical dysplasia/High Grade Squamous Intraepithelial Lesion with features for invasion (Reproductive system and breast disorders) | 0 (0) | 1 (1) — HPV16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clindamycin Phosphate Vaginal Gel, 2% (N=203) | Placebo Vaginal Gel (Universal HEC Placebo Gel) (N=103)
Vulvovaginal candidiasis (Infections and infestations) | 35 (37) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bacterial Vaginosis (Infections and infestations) | 3 (3) | 3 (3)
Bacterial vulvovaginitis (Infections and infestations) | 0 (0) | 1 (2)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Genital herpes (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Papilloma viral infection (Infections and infestations) | 0 (0) | 1 (1)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Trichomoniasis (Infections and infestations) | 4 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 6 (6) | 5 (5)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (2)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood pressure incrased (Investigations) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0)
Anosmia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervical friability (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervix disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 5 (5) | 4 (4)
Vulva cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulval disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Vulvovaginal erythema (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 9 (10) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT04370548/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT04370548/SAP_001.pdf